CLINICAL TRIAL: NCT01557855
Title: Enhanced Assessment of Chest Pain and Related Symptoms in the Primary Care Setting Through the Use of a Novel Personalized Medicine Genomic Test: Results From a Prospective Registry Study.
Brief Title: Investigation of a Novel Gene Expression Test (ASGES or Corus CAD) for Diagnosis of Obstructive Coronary Artery Disease
Acronym: REGISTRY-I
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000013; REGISTRY-I (Other: CardioDx)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Clinical Utility; Registry; Coronary Artery Disease; Coronary Heart Disease; Cardiovascular Disease; Angina Pectoris; Chest Pain; Registry I; Registry-I
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
The objective of this study is to collect data on the commercial use of Corus CAD (Age/Sex/Gene Expression score - ASGES) blood test to evaluate the clinical referral patterns of Primary Care Physicians after receipt of their patients' Corus Score, and to better understand patient management patterns for clinicians ordering the test.

DETAILED DESCRIPTION:
This is a prospective, multicenter observational registry collecting and analyzing commercial utilization data of the Corus CAD assay ("Test") also known as Age/Sex/Gene Expression score (ASGES) . The study will prospectively enroll approximately 670 evaluable subjects from qualified sites and evaluate the rate of referral versus Corus CAD (ASGES) score as continuous variables.

Objective of the study is to assess whether the score provided by the Corus CAD (Age/Sex/Gene Expression score - ASGES) test has an effect on the Primary Care Physician's patient management and referral patterns once received:

1. No further cardiac testing or treatment
2. Medical therapy for angina or non-cardiac chest pain
3. Referral to a cardiologist for stress testing with or without imaging, CT angiography, or invasive cardiac catheterization.

Since it takes approximately two days for the physician to receive the result of the Corus CAD (Age/Sex/Gene Expression score - ASGES) , initial diagnostic testing will reflect local standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms suggestive of CAD, including typical or atypical angina or angina equivalent
2. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form

Exclusion Criteria:

1. History of myocardial infarction
2. Current MI or acute coronary syndrome
3. Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms
4. Any previous coronary Revascularization
5. Any individuals with:

   * Diabetes
   * Suspected unstable angina
   * Systemic infections
   * Systemic inflammatory conditions
6. Any individuals currently taking:

   * Steroids
   * Immunosuppressive agents
   * Chemotherapeutic agents
7. Recipient of any organ transplant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled at multiple qualified participating study centers that have incorporated Corus CAD (ASGES) for the diagnosis of obstructive CAD into their routine practice.
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate of referral vs. Corus CAD (ASGES) score as continuous variables | 30 Days
  Composite endpoint consisting of referrals to a cardiologist, to cardiac stress/CTA and/or to invasive cardiac catheterization occurring between Day 0 and Day 30 + 15 days.

SECONDARY OUTCOMES:
Rate of referral difference between low Corus CAD or ASGES (</=15) and non-low ASGES (>15) scores. | 30 Day
  composite endpoint consisting of referrals to a cardiologist, to cardiac stress/CTA, and/or referral to invasive cardiac catheterization at Day 30 +15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, Study Director — CardioDx
Locations (7):
- United States (7):
  - Arizona Sun Family Medicine, Gilbert, Arizona
  - Fiel Family Medicine, Tempe, Arizona
  - Town Lake Internal Medicine, Woodstock, Georgia
  - Maringouin Medical Center, Maringouin, Louisiana
  - The Bonin Clinic, Zachary, Louisiana
  - Triangle Primary Care, Wake Forest, North Carolina
  - Comprehensive Physicians Associates, Youngstown, Ohio

REFERENCES:
- [Result] Ladapo JA, Lyons H, Yau M, Rich P, Newton D, Bruce-Mensah K, Johnson A, Zhou Y, Stemkowski S, Monane M. Enhanced assessment of chest pain and related symptoms in the primary care setting through the use of a novel personalized medicine genomic test: results from a prospective registry study. Am J Med Qual. 2015 Jul-Aug;30(4):345-52. doi: 10.1177/1062860614532517. Epub 2014 May 5. PMID 24798176
- [Derived] Ladapo JA, Herman L, Weiner BH, Rhees B, Castle L, Monane M, McPherson JA. Use of a blood test incorporating age, sex, and gene expression influences medical decision-making in the evaluation of women presenting with symptoms suggestive of obstructive coronary artery disease: summary results from two ambulatory care studies in primary care. Menopause. 2015 Nov;22(11):1224-30. doi: 10.1097/GME.0000000000000443. PMID 25828395